CLINICAL TRIAL: NCT01780064
Title: Active Early Individualized Psychosocial Accompaniment to Facilitate the Return to Employment of Women With Breast Cancer
Brief Title: Psychosocial Support to Facilitate the Return to Employment of Women With Breast Cancer
Acronym: APAPI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APAPI-1202
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard group (Placebo Comparator): routine monitoring with questionnaires
  Interventions: Behavioral: Questionnaires
- Interviews with psychologist (Active Comparator): Patients have interviews with a psychologist (at cure one of chemotherapy treatment,at cure six of chemotherapy treatment, at last radiotherapy session, and three months after the end of radiotherapy) and questionnaires
  Interventions: Behavioral: interviews with a psychologist; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: interviews with a psychologist — interviews with a psychologist
  Arms: Interviews with psychologist
Behavioral: Questionnaires — Questionnaires

SUMMARY:
The purpose of this study is to compare the effect of early individualized psychosocial assets versus a standard support on social inequalities in the rate of return to work

DETAILED DESCRIPTION:
For the group "intervention", patients have four interviews with a psychologist (at cure one of chemotherapy treatment, at cure six of chemotherapy treatment, at last radiotherapy session, and three months after the end of radiotherapy).

In the 2 arms, patients receive 4 sets of questionnaires (baseline, month 12, month 18 and month 24)

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 with work at the time of diagnosis
* Presenting a unilateral breast cancer exclusively local extension
* Having received surgery
* Reporting of adjuvant chemotherapy (+ / - trastuzumab)
* Reporting to radiotherapy or not (If radiotherapy, it will be done on site investigator)
* In work at the time of diagnosis (employees, traders and professionals)
* Patient affiliated to a social security scheme
* Consent signed by the patient before the implementation of any specific procedure to study

Exclusion Criteria:

* Presence of in situ lesions, cancer recurrence, metastatic disease immediately, location bilateral
* Inability physical, psychological, psychiatric or cognitive responses to the questionnaires and participate in interviews
* Recognition previous ALD (due to another disease)
* Patient under guardianship

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of early individualized psychosocial assets versus a standard support on social inequalities in the rate of return to work | At 24 months

SECONDARY OUTCOMES:
Comparison between the two modes of care, of social inequalities: | At 24 months
  * On the quality of the return to employment (working conditions, job stability)
  * On individual and collective resources of patients (social encouragement received, reactions to issues, anxiety/depression, quality of life, etc)
Calculating the cost / benefit ratio of the two modes of care | At 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie FANTONI, MD, PhD, Study Director — CHRU / Université Lille 2; Jacques BONNETERRE, MD, PhD, Study Director — Centre Oscar Lambret
Locations (7):
- France (7):
  - Centre Marie Curie, Arras
  - Centre Pierre Curie, Beuvry
  - Centre Léonard de Vinci, Dechy
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier, Valenciennes
  - Nouvelle Clinique des Dentellières, Valenciennes
  - Hôpital Privé de Villeneuve d'Ascq, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No